CLINICAL TRIAL: NCT03581578
Title: VITROS Immunodiagnostic Products hs Troponin I
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ortho-Clinical Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-002
Record Dates: First submitted 2018-04-19; First posted 2018-07-10 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Acute Coronary Syndrome (ACS); Myocardial Infarction
Keywords: Troponin
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Prospective collection of serial blood samples with serum and lithium heparin plasma.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this clinical study is to collect data to substantiate the use of the VITROS hs Troponin I test as an aid in the diagnosis of myocardial infarction (MI). The test is further indicated for risk stratification of mortality, myocardial infarction or coronary revascularization in patients with acute coronary syndrome.

DETAILED DESCRIPTION:
A prospective clinical sample collection and cardiac troponin I testing will be conducted in individuals presenting to the Emergency Department (ED) with signs and/or symptoms suggestive of acute coronary syndrome (ACS) at geographically dispersed sites in the US. Individuals who meet the inclusion/exclusion criteria, including having signed an informed consent form will be included in the study.

Clinical and laboratory data will be collected to demonstrate product performance compared to an adjudicated clinical diagnosis.

Sample collection and testing of clinical samples with the VITROS hs Troponin I test will be performed under two separate protocols.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥22 years of age at the time of consent.
2. Subject presenting with symptoms suggestive of acute coronary syndrome including chest pain, or chest pain equivalent.
3. Must have an Electrocardiogram (ECG) ordered as part of the subject's standard of care.
4. Subject willing and able to provide informed consent.

Exclusion Criteria:

1. Subject is unable to comply with the study requirements.
2. Any samples which were not obtained under IRB approved protocol.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals presenting to the Emergency Department (ED) with signs and/or symptoms suggestive of acute coronary syndrome (ACS).
Sampling Method: Non-Probability Sample
Enrollment: 1630 (Estimated)
Dates: Start 2018-06-07 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the VITROS hs Troponin I test | VITROS hs Troponin I value at baseline
  Evaluate the sensitivity and specificity of the VITROS hs Troponin I test result against the adjudicated diagnosis for subjects with acute coronary syndrome (ACS).
Sensitivity and specificity of the VITROS hs Troponin I test | VITROS hs Troponin I value > 1 hour and up to 3 hours
  Evaluate the sensitivity and specificity of the VITROS hs Troponin I test result against the adjudicated diagnosis for subjects with acute coronary syndrome (ACS).
Sensitivity and specificity of the VITROS hs Troponin I test | VITROS hs Troponin I value at > 3 hours and up to 6 hours
  Evaluate the sensitivity and specificity of the VITROS hs Troponin I test result against the adjudicated diagnosis for subjects with acute coronary syndrome (ACS).
Sensitivity and specificity of the VITROS hs Troponin I test | VITROS hs Troponin I value at > 6 hours and up to 9 hours
  Evaluate the sensitivity and specificity of the VITROS hs Troponin I test result against the adjudicated diagnosis for subjects with acute coronary syndrome (ACS).

SECONDARY OUTCOMES:
Risk stratification of subjects | Up to 12 months after last enrollment
  Assess the use of cardiac Troponin I measurement in the risk stratification of subjects.
Rule in and rule out myocardial infarction (MI) | VITROS hs Troponin I values from two collection time points (baseline, > 1 hour and up to 2 hours)
  Evaluate the VITROS hs Troponin I test to rule in and rule out MI.

CONTACTS AND LOCATIONS:
Overall Officials: Fred Apple, PhD, Principal Investigator — Hennepin Healthcare Research Institute; Richard Nowak, MD, Principal Investigator — Henry Ford Health System
Locations (24):
- United States (24):
  - Drug Research and Analysis Corp, Montgomery, Alabama
  - Chandler Regional Medical Center, Chandler, Arizona
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Maryland, Baltimore, Maryland
  - Mass General Hospital, Boston, Massachusetts
  - Wayne State University/Detroit Receiving Hospital, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Beaumont, Royal Oak, Michigan
  - Hennepin County Medical Center/Minneapolis Medical Research Foundation, Minneapolis, Minnesota
  - Cooper University Hospital, Camden, New Jersey
  - Stony Brook University Hospital, Stony Brook, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Oregon Health Science University Hospital, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Tech University Health Sciences Center El Paso, El Paso, Texas
  - Ben Taub General Hospital / Baylor College of Medicine/Harris Health System, Houston, Texas
  - INOVA Alexandria Hospital, Alexandria, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Charleston Area Medical Center, Charleston, West Virginia
  - Medical College of Wisconsin and Froedtert Hospital, Milwaukee, Wisconsin